CLINICAL TRIAL: NCT04521998
Title: Comparative Effectiveness Research of Electroacupuncture and Transcutaneous Electrical Nerve Stimulation in Patients With Rheumatoid Arthritis: A Pragmatic Randomized Clinical Trial
Brief Title: Comparative Effectiveness Research of Electroacupuncture and TENS in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC1-100
Record Dates: First submitted 2020-08-16; First posted 2020-08-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: Comparative effectiveness research; electroacupuncture; transcutaneous electrical nerve stimulation; rheumatoid arthritis:; randomized clinical trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Electroacupuncture; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Experimental): The needles remained in situ for 30 minutes, during which time the acupuncturist returned to stimulate the needles once to re-elicit the de qi sensation. Participants have 2 sessions per week, with total 5 weeks and 10 sessions. The body points included LI4, LI11, SP6 and ST36. The individual specific points protocol are as follows: GB20, TE5, SP10, GB34, LV3, ba xie, ba fen, Ashi). The acupuncture protocol consists of the body points and some of the individual specific points depending on subjects' condition.
  Interventions: Device: electroacupuncture
- Transcutaneous electrical nerve stimulation (Experimental): The protocol consisted of first swabbing all points with alcohol, then pads of TENS were sticked on the proper location of acupoints included LI4, LI11, SP6 and ST36. Electrical output of one channel was administered to the surface of body via a combination of two pads. LI4 and LI11, ST36 and SP6 are combination of acupoints, respectively. Participants had 2 sessions per week, with total 5 weeks and 10 sessions. Each session lasted 30 minutes.
  Interventions: Device: TENS

INTERVENTIONS:
Device: electroacupuncture — Electroacupuncture used to reduce the inflammation was proved previously.
  Arms: electroacupuncture
Device: TENS — Patients who unlike needles would like to choose TENS as treatment for pain relief.
  Arms: Transcutaneous electrical nerve stimulation

SUMMARY:
The aim of this pilot study is to compare the effectiveness of electroacupuncture or transcutaneous electrical nerve stimulation in reducing the tenderness in the patients with rheumatoid arthritis. The study adopted a pragmatic, randomized, patient-centered approach to investigate the effectiveness of clinical symptoms and quality of life.

DETAILED DESCRIPTION:
A total of 80 volunteers of patients with rheumatoid arthritis will be recruited from the Chinese medicine or Western medicine clinics in China Medical University Hospital and Dalin Tzu-Chi Hospital. These patients will be randomized to receive electroacupuncture (40 participants) or transcutaneous electrical nerve stimulation (40 participants) treatment two sessions per week and for 10 treatments in total.

The investigators expect that electroacupuncture or transcutaneous electrical nerve stimulation can reduce the severity of pain in the patients with rheumatoid arthritis. The effectiveness of electroacupuncture or transcutaneous electrical nerve stimulation can be detected by visual analogue scale, simplified disease activity index, and disease activity score and be used to improve the clinical symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old
* Met the American College of Rheumatology criteria (2010) for RA
* Classification of X-ray : Stage I~III
* The participants' RA medication regimen (DMARD, NSAID, steroid)were eligible if they were on a stable dose for at least 3 months before entry into and throughout the study.
* All patients were instructed not to make any changes in their background therapies during the study.
* Intra-articular or pulse steroid were not permitted during the study

Exclusion Criteria:

* Be treated with biological agents, such as antagonist of TNF-alpha, IL-6, Jak, and CD20 mono antibody in the last 3 months
* Having history of serious drug allergy
* Pregnancy or breastfeeding
* Bleeding or coagulation disorders
* Localized skin infections
* Uncontrolled or ill-controlled blood pressure with diastolic pressure≥110 mmHg
* Any other acupuncture treatment or herbal medication for RA within 2 weeks before screening
* needle phobia
* Intra-articular corticosteroid or pulse steroid within 4 weeks preceding the study
* Any severe chronic or uncontrolled comorbid disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Morning stiffness(scoring range 0~10 and lasting time : min/day) | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed

SECONDARY OUTCOMES:
Simplified disease activity index (scoring range 0.0 ~ 86.0) | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed
Disease Activity Score 28 (scoring range 0.0 ~ 9.4) | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed
Erythrocyte sedimentation rate | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed
Clinical Disease Activity Index (scoring range 0.0 ~ 76.0) | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed
Pain Visual Analogue Scale (scoring range 0 ~ 10) | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed
C-reactive protein | baseline, week 5, and week 9
  Changes from baseline to end of intervention and 4 weeks after intervention completed

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, M.D. Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No